CLINICAL TRIAL: NCT01627327
Title: A 12-Week Study to Evaluate the 24-Hour Pulmonary Function Profile of Fluticasone Furoate /Vilanterol (FF/VI) Inhalation Powder 100/25mcg Once-Daily Via a Novel Dry Powder Inhaler Compared With Tiotropium Bromide Inhalation Powder 18mcg Delivered Once-Daily Via the HandiHaler in Subjects With Chronic Obstructive Pulmonary Disease (COPD) Who Have or Are at Risk for Co-morbid Cardiovascular Disease
Brief Title: Study to Evaluate the 24-Hour Pulmonary Function Profile of Fluticasone Furoate/Vilanterol (FF/VI) Inhalation Powder 100/25mcg Once Daily Compared With Tiotropium Bromide Inhalation Powder 18mcg Once Daily in Subjects With COPD Who Have or Are At Risk for Co-morbid Cardiovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115805
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Cardiovascular event; Cardiovascular disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases | interventions — fluticasone furoate; vilanterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone furoate/vilanterol (Experimental): inhaled corticosteroid (ICS)/long-acting beta2-agonist (LABA)
  Interventions: Drug: fluticasone furoate/vilanterol 100/25mcg
- tiotropium bromide (Active Comparator): anticholinergic
  Interventions: Drug: tiotropium bromide 18mcg

INTERVENTIONS:
Drug: fluticasone furoate/vilanterol 100/25mcg — inhalation powder
  Arms: fluticasone furoate/vilanterol
Drug: tiotropium bromide 18mcg — inhalation powder
  Other Names: Spiriva
  Arms: tiotropium bromide

SUMMARY:
The purpose of this study is to evaluate the 24-hour spirometry effect (FEV1) of Fluticasone Furoate/Vilanterol Inhalation Powder 100/25mcg once daily compared with tiotropium bromide inhalation powder 18mcg once daily over a 12-week treatment period in subjects with COPD who have or are at risk for co-morbid cardiovascular disease

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, multi-center, parallel-group study. Subjects who meet the eligibility criteria at Screening and at the end of a 2-week Run-In Period will enter a 12-week Treatment Period. There will be a 7-day Follow-up Period after the Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Male or females ≥ 40 years of age
* Females must be post-menopausal or using a highly effective method for avoidance of pregnancy
* Established clinical history of COPD by ATS/ERS definition
* Post-albuterol spirometry criteria: FEV1/FVC ratio ≤ 0.70 and FEV1 ≥30 to ≤ 70% of predicted normal (NHANES III)
* Former or current smoker ≥10 pack years
* A history of diagnosed cardiovascular disease or a prior cardiovascular event including any of the following:
* Established (i.e., by clinical signs or imaging studies) coronary artery disease (CAD)
* Established (i.e., by clinical signs or imaging studies) peripheral vascular (i.e., arterial) disease (PVD)
* Previous stroke
* Objectively confirmed transient ischemic attack (TIA) (i.e., transient neurological deficit documented by a health-care professional)
* Previous myocardial infarction (MI) (Note: An MI within 6 months prior to Visit 1 is exclusionary)

OR

* Presence of one of the following cardiovascular risk factors (in addition to being a former/current smoker):
* Current diagnosis of hypertension
* Current diagnosis of hypercholesterolemia
* Diabetes mellitus treated with pharmacotherapy

Exclusion Criteria:

* Current diagnosis of asthma
* Subjects with other respiratory disorders including α1-antitrypsin deficiency as the underlying cause of COPD, active tuberculosis, lung cancer, bronchiectasis (Note: focal bronchiectasis is not exclusionary), sarcoidosis, pulmonary fibrosis (Note: focal fibrotic pulmonary lesions are not exclusionary), pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
* Lung volume reduction surgery within previous 12 months
* Clinically significant abnormalities not due to COPD by chest X-ray or CT scan
* Hospitalized for poorly controlled COPD within 12 weeks of Screening
* Poorly controlled COPD 6 weeks prior to Screening, defined as acute worsening of COPD that is managed by the subject with corticosteroids or antibiotics or that requires treatment prescribed by a physician
* Lower respiratory infection requiring antibiotics 6 weeks prior to Screening
* A moderate or severe COPD exacerbation and/or a lower respiratory tract infection (including pnuemonia) during the Run-In Period
* An abnormal, clinically significant finding in any liver chemistry, biochemical, or haematology tests at Screening (Visit 1) or upon repeat prior to randomization
* An abnormal, clinically significant ECG finding at Screening (Visit 1) or upon repeat prior to randomization
* An abnormal, clinically significant Holter finding at Screening (Visit 1) or upon repeat prior to randomization (sub-set of subjects)
* Historical or current evidence of clinically significant (in opinion of the Investigator) and unstable disease such as cardiovascular (e.g., patients requiring ICD, pacemaker requiring a ventricular pace rate set at >60 bpm, uncontrolled hypertension, New York Heart Association Class IV (New York Heart Association,1994), known left ventricular ejection fraction <30%), neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease), peptic ulcer disease, or haematological abnormalities
* Carcinoma not in complete remission for at least 5 years
* History of allergy or hypersensitivity to any of the study medications (e.g., anticholinergic/muscarinic receptor antagonist, beta2-agonist, corticosteroid) or components of the inhalation powder (e.g., lactose, magnesium stearate) or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic. In addition, subjects with a history of severe milk protein allergy that, in the opinion of the Investigator, contraindicates the subject's participation will also be excluded
* Known/suspected history of alcohol or drug abuse in the last 2 years
* Women who are pregnant or lactating or plan to become pregnant
* Subjects medically unable to withhold albuterol /salbutamol for 4 hours prior to spirometry testing at each study visit
* Use of certain medications such as bronchodilators and corticosteroids for the protocol-specific times prior to Visit 1 (the Investigator will discuss the specific medications)
* Long Term Oxygen Therapy (LTOT) or nocturnal oxygen therapy >12 hours a day
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Screening or during the study
* Failure to demonstrate adequate compliance defined as completion of the Diary Card (completed all diary entries on at least 4 of the last 7 consecutive days), the ability to withhold COPD medications and to keep clinic visit appointments
* Non-compliance or inability to comply with study procedures or scheduled visits
* History of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study
* Affiliation with investigator site
* Women who are pregnant or lactating or are planning on becoming pregnant during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2012-04-01; Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (11):
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Newport News, Virginia
- Canada (7):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Czechia (5):
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Kroměříž
  - GSK Investigational Site, Teplice
  - GSK Investigational Site, Třebíč
  - GSK Investigational Site, Žamberk
- Germany (10):
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Poland (7):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Działdowo
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Piekary Śląskie
  - GSK Investigational Site, Słupsk
  - GSK Investigational Site, Tarnów
- Romania (6):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 115805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115805 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants (par.) completed a 2-week Run-in Period (RIP) to obtain baseline assessments of rescue use, COPD symptom scores and disease stability. Par. were then randomized to a 12-week Treatment Period. A total of 890 par. were screened, of whom 623 were randomized and received at least one dose of study medication.
Groups:
- FF/VI 100/25 µg OD: Participants received Fluticasone Furoate /Vilanterol (FF/VI) 100/25 micrograms (µg) inhalation once daily (OD) via a dry powder inhaler (DPI) and placebo inhalation OD via a HandiHaler in the morning for 12 weeks.
- TIO 18 µg OD: Participants received tiotropium bromide (TIO) 18 µg inhalation OD via a HandiHaler and placebo inhalation OD via a DPI in the morning for 12 weeks.
Period: Overall Study
Arm/Group | FF/VI 100/25 µg OD | TIO 18 µg OD
Started | 310 | 313
Completed | 291 | 274
Not Completed | 19 | 39
Not completed — Adverse Event | 6 | 12
Not completed — Lack of Efficacy-No Sub-Reason | 0 | 2
Not completed — Lack of Efficacy-Sub-Reason Exacerbation | 4 | 9
Not completed — Protocol Violation | 4 | 10
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- FF/VI 100/25 µg OD: Participants received FF/VI 100/25 µg inhalation OD via a DPI and placebo inhalation OD via a HandiHaler in the morning for 12 weeks.
- TIO 18 µg OD: Participants received TIO 18 µg inhalation OD via a HandiHaler and placebo inhalation OD via a DPI in the morning for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | FF/VI 100/25 µg OD | TIO 18 µg OD | Total
Number analyzed (Participants) | 310 | 313 | 623
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (8.09) | 62.3 (7.98) | 62.6 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 104 | 221
  Male | 193 | 209 | 402
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 8 | 7 | 15
  Asian - East Asian Heritage | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 302 | 305 | 607

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Trough in 24-hour Weighted Mean FEV1 on Treatment Day 84
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled from the lungs in one second. The weighted mean was calculated from the pre-dose FEV1 and post-dose FEV1 measurements at 5, 15, 30 minutes and 1, 2, 4, 6, 8, 12, 13, 14, 16, 20, and 24 hours on Treatment Day 84. Baseline trough FEV1 was the mean of the two assessments made 30 and 5 minutes pre-dose on Treatment Day 1. Change from Baseline (BL) was calculated as the average of the Day 84 values minus the Baseline value. Analysis was performed using an analysis of covariance (ANCOVA) model with covariates of BL FEV1, exacerbation history and reversibility stratum, smoking status at screening, country, and treatment group.
Time Frame: Baseline and Day 84
Population: Intent-to-Treat (ITT) Population: all participants who were randomized and received at least one dose of study medication. Only participants with data available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF/VI 100/25 µg OD | TIO 18 µg OD
Number analyzed (Participants) | 254 | 236
Liters | 0.117 (0.0130) | 0.095 (0.0138)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg OD vs TIO 18 µg OD; Test type: Superiority or Other; p = 0.201, ANCOVA; Median Difference (Net) = 0.022, 95% CI 2-sided [-0.012 to 0.055]

2. Secondary Outcome: Time to Onset on Treatment Day 1
Description: Time to onset on Treatment Day 1 is defined as the time to an increase of 100 milliliters (mL) from Baseline in FEV1. Time of onset was calculated over 0 to 4 hours (5 minutes (min), 15 min, 30 min, 60 min, 120 min, and 240 min) post-dose. Time to onset was analyzed using a log-rank test, stratified by exacerbation history and reversibility stratum.
Time Frame: Baseline and Day 1
Population: ITT Population. Only participants with data available at the indicated time point were assessed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | FF/VI 100/25 µg OD | TIO 18 µg OD
Number analyzed (Participants) | 239 | 254
Minutes | 17.0 [5 to 240] | 20.5 [5 to 240]

3. Secondary Outcome: Change From Baseline in Trough FEV1 at Treatment Day 84
Description: Pulmonary function was measured by FEV1. Trough FEV1 was defined as the 24-hour FEV1 assessment, which was obtained on Day 84. Baseline is defined as the mean of the two assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1.Change from Baseline was calculated as the average of the Day 84 values minus the Baseline value. Analysis was performed using an ANCOVA model with covariates of BL FEV1, exacerbation history and reversibility stratum, smoking status at screening, country, and treatment group.
Time Frame: Baseline and Day 84
Population: ITT Population. Only participants with data available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF/VI 100/25 µg OD | TIO 18 µg OD
Number analyzed (Participants) | 268 | 249
Liters | 0.098 (0.0133) | 0.093 (0.0140)

ADVERSE EVENTS:
Time Frame: On-Treatment serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until Follow-up (up to 13 weeks).
Description: An on-treatment AE or SAE is defined as an AE with an onset on or after the start date of study medication, but not later than one day after the last date of study medication. SAEs and AEs were collected in members of the ITT Population, comprised of all participants randomized to treatment, who received at least one dose of study medication.
Arm/Group | FF/VI 100/25 µg OD | TIO 18 µg OD
Serious Adverse Events (participants affected / at risk) | 10/310 | 10/313
Other Adverse Events (participants affected / at risk) | 31/310 | 32/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg OD (N=310) | TIO 18 µg OD (N=313)
Pneumonia (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Graft infection (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 1 | 0
Leriche syndrome (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg OD (N=310) | TIO 18 µg OD (N=313)
Headache (Nervous system disorders) | 18 | 23
Nasopharyngitis (Infections and infestations) | 16 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.